CLINICAL TRIAL: NCT07080827
Title: The Effect of Transtheoretical Model-Based Psychoeducation Via Social Media on Treatment Adherence in Individuals Diagnosed With Psychosis
Brief Title: TTM-Based Social Media Psychoeducation for Psychosis
Acronym: TAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ibrahim Aldemir, PhD, Doctoral Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024229
Record Dates: First submitted 2025-07-11; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Treatment Compliance; Social Media; Psychotic Disorders
Keywords: Treatment Compliance and Compliance; Mental Health Nursing; Online Psychoeducation
MeSH Terms: conditions — Patient Compliance; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online TTM-Based Psychoeducation (Experimental)
  Interventions: Behavioral: TTM-Based Online Psychoeducation Program
- Face-to-Face Standard Psychoeducation (Active Comparator)
  Interventions: Behavioral: Standard Face-to-Face Psychoeducation Program
- Delayed Online Psychoeducation Group (Active Comparator)
  Interventions: Other: TTM-Based Online Psychoeducation Program

INTERVENTIONS:
Behavioral: TTM-Based Online Psychoeducation Program — A 5-week structured psychoeducation program based on the Transtheoretical Model (TTM), delivered via WhatsApp. Educational content was tailored to the participant's stage of change and included videos, texts, and interactive materials to promote treatment adherence in individuals with psychosis.
  Arms: Online TTM-Based Psychoeducation
Behavioral: Standard Face-to-Face Psychoeducation Program — A 3-week conventional psychoeducation program delivered face-to-face at the Community Mental Health Center. The program focused on general treatment adherence without utilizing the Transtheoretical Model and included verbal education, printed materials, and discussions.
  Arms: Face-to-Face Standard Psychoeducation
Other: TTM-Based Online Psychoeducation Program — The intervention was provided after a 3-month delay following initial observation. Participants received the same 5-week online psychoeducation program as the main intervention group
  Arms: Delayed Online Psychoeducation Group

SUMMARY:
This doctoral research investigates the effect of a Transtheoretical Model (TTM)-based psychoeducation program delivered via social media on treatment adherence in individuals diagnosed with psychosis. The study follows a randomized controlled trial design with pretest, posttest, and three-month follow-up assessments.

A total of 60 participants were selected from among 354 individuals registered at the Balıkesir Community Mental Health Center (CMHC), based on predefined inclusion and exclusion criteria. Participants were randomly assigned into three groups:

1. an online intervention group receiving a 5-week TTM-based treatment adherence psychoeducation program via WhatsApp;
2. a face-to-face intervention group receiving a standard, non-TTM-based treatment adherence psychoeducation program over 3 weeks at the CMHC; and
3. a control group that received no educational intervention, only assessments.

Data collection instruments include a Sociodemographic Information Form, the Stage of Change Identification Form, the Medication Adherence Report Scale (MARS-5), and the Clinical Global Impression-Severity Scale (CGI-S). Measurements were conducted at baseline, post-intervention, and three months after the intervention.

The study hypotheses are:

Research Hypotheses H1: The treatment adherence scale scores of individuals diagnosed with psychosis who participate in the TTM-based psychoeducation group administered via social media will differ compared to the scores of individuals who participate in the face-to-face treatment adherence psychoeducation group.

H2: The treatment adherence scale scores of individuals diagnosed with psychosis who participate in the TTM-based psychoeducation group administered via social media will differ compared to the scores of individuals who do not receive TTM-based psychoeducation.

This study aims to provide evidence for the efficacy of theory-based, technology-supported psychoeducation programs in enhancing treatment adherence among individuals with psychosis. Furthermore, it evaluates whether a model-based online psychoeducation program is more effective than a conventional treatment adherence education.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosed with a psychotic disorder according to DSM-5 criteria, including:
* Schizophrenia
* Schizophreniform disorder
* Schizoaffective disorder (with mild mood symptoms)
* Brief psychotic disorder
* Substance/medication-induced psychotic disorder (in remission)
* Paranoid disorder
* On the same prescribed psychiatric medication for at least one month
* Able to communicate in Turkish
* Has access to the internet and owns at least one active social media account (Instagram, Twitter, Facebook, WhatsApp, etc.)
* Literate and able to complete self-report forms
* Willing to participate and provide informed consent
* Clinical Global Impression-Severity (CGI-S) score of 4 or below

Exclusion Criteria:

* Under 18 or over 65 years of age
* Acute psychotic episode at the time of recruitment
* Comorbid psychiatric diagnoses not covered under the inclusion list
* Diagnosed with neurocognitive disorders (e.g., dementia)
* Diagnosed with intellectual disability (mental retardation)
* Unable to use smartphone, tablet, or other digital communication tools
* Missed more than 20% of the intervention sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence (Treatment adherence) | Baseline (Week 0) and Post-Intervention (Week 5)
  Score on a 5-point Likert scale
Change in Medication Adherence Scores (MARS-5) | Baseline, Post-Intervention (Week 5), and 3-Month Follow-Up
  Medication adherence will be assessed using the 5-item Medication Adherence Report Scale (MARS-5), originally developed by Horne and Hankins (2001). It is a generic, self-reported Likert-type scale validated across various chronic physical and psychiatric conditions, including bipolar disorder, hypertension, asthma, and schizophrenia. Each item is rated on a 5-point scale from 1 (always) to 5 (never), yielding a total score between 5 and 25. Higher scores indicate better adherence.
  The Turkish version of the scale was adapted by the investigators and demonstrated acceptable internal consistency (Cronbach's α = 0.78). Factor analyses supported a unidimensional structure (KMO = 0.79; CFI = 0.97; RMSEA = 0.089), consistent with the original.
  In this study, MARS-5 will be administered at three time points: prior to the intervention (baseline), immediately following the intervention (post-test), and three months after the intervention (follow-up) to assess changes in treatment adherence

CONTACTS AND LOCATIONS:
Locations (1):
- Balıkesir Provincial Health Directorate, Community Mental Health Center, Balıkesir, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No